CLINICAL TRIAL: NCT00098046
Title: Pharmacokinetics and Safety of Famciclovir Oral Pediatric Formulation in Children 1-12 Years of Age With Varicella Zoster Infection
Brief Title: Famciclovir Oral Pediatric Formulation in Children 1-12 Years of Age With Varicella Zoster Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFAM810B2304
Record Dates: First submitted 2004-12-02; First posted 2004-12-03 (Estimated); Last update posted 2007-09-26 (Estimated); Status verified 2007-09

CONDITIONS: Chickenpox; Herpes Zoster
Keywords: chickenpox; herpes zoster; children; Famvir; varicella zoster virus
MeSH Terms: conditions — Chickenpox; Herpes Zoster | interventions — Famciclovir

INTERVENTIONS:
Drug: famciclovir

SUMMARY:
Varicella zoster virus causes chickenpox in children and shingles in adults. Chickenpox is usually a self-limiting illness characterized by fever and a rash. Serious complications can include secondary bacterial infections, pneumonia, and encephalitis. Anti-viral treatment is not a standard of care in immunocompetent children, but is recommended whenever a risk of complication exists. This study will evaluate the safety and blood levels of a new formulation of famciclovir in children 1-12 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Male or female children 1-12 years of age
* Clinical or laboratory evidence of varicella zoster infection
* Patients suspected of having varicella zoster infection

Exclusion Criteria:

* Patients unable to swallow
* Concomitant use of probenecid
* Positive pregnancy

Additional protocol-defined inclusion/exclusion criterial may apply. For detailed information on eligibility, please contact the study center nearest to you (see below), or call the following number 1-862-778-3544 or 1-434-951-3228

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Estimated)
Dates: Start 2005-07; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Step A: Single-dose safety and pharmacokinetics
Step B: Safety and tolerability of pediatric formulation administered 3 times daily over 7 days

SECONDARY OUTCOMES:
Steps A & B: Acceptability of pediatric formulation by patients

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (5):
- Columbia University Medical Center, New York, New York, United States
- Novartis Investigational Site, San José, Costa Rica
- Novartis Investigational Site, Cuidad de Guatemala, Guatemala
- Panama (2):
  - Novartis Investigational Site, David, Chiriqui
  - Novartis Investigational Site, Panama City

REFERENCES:
- [Derived] Saez-Llorens X, Yogev R, Arguedas A, Rodriguez A, Spigarelli MG, De Leon Castrejon T, Bomgaars L, Roberts M, Abrams B, Zhou W, Looby M, Kaiser G, Hamed K. Pharmacokinetics and safety of famciclovir in children with herpes simplex or varicella-zoster virus infection. Antimicrob Agents Chemother. 2009 May;53(5):1912-20. doi: 10.1128/AAC.01054-08. Epub 2009 Mar 9. PMID 19273678